CLINICAL TRIAL: NCT05450640
Title: Evaluation of the Evolution of the Patient Care Pathway in the Context of the Implementation of the DOuBLE EMIcizumab Dispensing Circuit in France
Brief Title: Satisfaction Regarding the Dispensing of Emicizumab (HEMLIBRA®) for Patients With Haemophilia A in France
Acronym: PASODOBLEDEMI2
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: PASODOBLEDEMI2
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Accessibility; Emicizumab (HEMLIBRA®); Patient satisfaction
MeSH Terms: conditions — Hemophilia A; Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with haemophilia A with dispensing Emicizumab (HEMLIBRA®) in community pharmacy: This group of patients have chosen the dispensing of Emicizumab (HEMLIBRA®) in community pharmacy. This choice involves the contribution of the community pharmacist in the dispensing circuit who does not replace the hospital pharmacist but interact together for prescriptions renewals, emergency treatment or sharing information if necessary.
  Interventions: Other: satisfaction survey
- Patients with haemophilia A with dispensing Emicizumab (HEMLIBRA®) in hospital pharmacy: This group of patients have kept the dispensing of Emicizumab (HEMLIBRA®) in hospital pharmacy
  Interventions: Other: satisfaction survey

INTERVENTIONS:
Other: satisfaction survey — 1 eQuestionnaire per patient completed during study

SUMMARY:
Haemophilia A (HA) is a rare constitutional haemorrhagic disease whose drug management is based on the use of chronic lifelong replacement therapy. The occurrence of an inhibitor is a dreaded complication that impacts conventional management, consisting in using factor VIII (FVIII)-based replacement therapy, most often for prophylaxis. Although effective, these treatments can only be administered intravenously, leading to accessibility constraints and significant mental burden for patients and their relatives.

Before June 15, 2021 in France, the emicizumab (HEMLIBRA®) was available only in hospital pharmacies for the prevention or reduction of bleedings. The introduction of the dual dispensing circuit in hospital or community pharmacies, left to patient's choice, is effective from this date. These changes have important organizational consequences for patients and health professionals alongside the pathway of care. Therefore, the effectiveness of this new organization requires to be evaluated with a national French study, called PASO DOBLE DEMI. The aims of this study are twofold :

I. To evaluate the direct impact of the training programs provided to the new placeholders of the dispensing circuit ; the community pharmacists, II. To evaluate satisfaction of patients or their relatives regarding the emicizumab treatment whether they chose dispensing in the community pharmacy, or kept the dispensing at the hospital pharmacy.

The methodology was based on the 4-level of the Kirkpatrick's evaluation model; 1) the immediate reaction of community pharmacists following the trainings (Reaction), 2) their knowledge acquisition (Learning), 3) their professional practice (Behavior) and 4 ) the patients' satisfaction related to their treatment whether dispensing in hospital or in community pharmacies (Results).

The PASO DOBLE DEMI II study was based on the fourth level of the evaluation model and particularly to evaluate to what extent the dispensing of Emicizumab (HEMLIBRA ®) treatment in community pharmacies has contributed to the improvement of the satisfaction of patients with HA.

The availability of the treatment in community pharmacy assumes an improvement of the treatment accessibility for the patient at several levels :

* Global accessibility: what choice has the patient expressed to access his treatment from a practical point of view?
* Adaptation: Has the patient adapted to the new treatment delivery organization?
* Availability of resources: are the special needs of the patients taken into consideration?
* Social acceptability: is the patient willing to follow the proposed care pathway? The issue of treatment cost is not considered in this study because the cost of antihemophilic treatments is totally covered by the French government for all patients regardless of their insurance coverage

ELIGIBILITY:
Inclusion Criteria:

* Patient with hemophilia type A with or without inhibitors
* Patients treated with Emicizumab (Hemlibra®)
* Age over 18 years old or legal representative of a minor haemophilia type A patient or his/her relative/caregiver for a non-autonomous adult patient

Exclusion Criteria:

* Patient under guardianship / curatorship
* Opposition expressed to use personal data

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: With approximately one in 6,000 men with haemophilia A, we estimated about 2,900 patients in France with 35% of cases with severe haemophilia, 15% of cases with moderate haemophilia and 50% of cases with minor severity. The eligible population for inclusion in the study considered all patients, regardless of age, treated with Emicizumab (HEMLIBRA®), whether they choose dispensing in community pharmacies, or retained dispensing in hospital pharmacy. The Laboratory Roche-Chugai which commercialize Emicizumab (HEMLIBRA®) estimated about 1'000 patients eligible to the inclusion criteria. We assumed that the uptake of the dispensing circuit, and therefore the number of patients choosing dispensing in community pharmacies, approximated the number of trained pharmacists.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-01-09 (Actual); Study Completion 2023-01-09 (Actual)

PRIMARY OUTCOMES:
satisfaction levels reported through a specific questionnaire | 6 months
  This questionnaire is composed of 40 questions for an estimated time to fulfil not exceeding 8 minutes. The overall satisfaction levels consists in collecting the patient's perception based on the 4-item of the Likert-scale (strongly dissatisfied, rather not satisfied, rather satisfied, strongly satisfied) taking into account the 4 dimensions of accessibility (global accessibility, adaptation, availability of resources, social acceptability).

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Chamouard, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fraticelli L, Freyssenge J, Prome-Combel E, Agnellet E, Dargaud Y, Chamouard V. Evaluation of the Care Pathway in the Context of the Dispensing of Emicizumab (Hemlibra) in Community Pharmacies in France: Protocol for a Cross-sectional Study Based on the Kirkpatrick Model. JMIR Res Protoc. 2023 Mar 8;12:e43091. doi: 10.2196/43091. PMID 36884286